CLINICAL TRIAL: NCT00946439
Title: Wheel Assisted Running Training in Children With Cerebral Palsy: A Controlled Clinical Trial
Brief Title: Wheel Assisted Running Training (WART) in Children With Cerebral Palsy
Acronym: WART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Israel Sport Center for the Disabled (Other)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Ziva Yizhar, Dept. Physical Therapy Faculty of Medicine Tel Aviv University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Revital123
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2009-07-27 (Estimated); Status verified 2009-07

CONDITIONS: Cerebral Palsy
Keywords: training exercise gait
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Wheel assisted running training — 'Race-Runner' uses the principle of body weight reduction and wheel assisted running training. This is a three-wheel device specifically designed in the 1990s for athletic purposes. The participant is walking or running with the feet on the ground while using a triangular frame equipped with three large bicycle wheels. Support to the participant's body is provided by a regular cycle saddle, a frontal body support plate, and the steering handlebars. The vertical and horizontal distance of the saddle and frontal support from the steering handlebars are adaptable to the participant's body dimension and comfort. This equipment is commonly used in competition in Scandinavia and Central Europe
  Other Names: also called 'Petra'

SUMMARY:
The purpose is to evaluate the effects of adding a wheel assisted running training (WART) to a conventional mixed physical activity training (CT) program on walking and gross motor function in trained children with cerebral palsy (CP).

Method entails recruiting thirty children with CP (16 females, 14 males), with mean (SD) age 11.8 (3.5) and training experience 3.4 (3.5), years were assigned to either WART or CT groups. The energy Expenditure Index (EEI), the Gross Motor Function Measure 66 (GMFM), self-selected and fast walking velocity (SSV and FV, respectively), and cadence are administered by a trained physical therapist. The intervention period is six months, with two sessions per week.

ELIGIBILITY:
Inclusion Criteria:

* (a) medical diagnosis of cerebral palsy;
* (b) ability to comprehend instructions in a group setting;
* (c) no medical procedures involving the lower limbs (including casting and Botox injections) during the last six months prior to pre-testing;
* (d) able to walk three minutes at a self paced speed;
* (e) no seizures during the last year, and (f) functional performance levels between II-IV of the gross motor functional classification system (GMFCS)

Exclusion Criteria:

* (a) GMFCS I or V;
* (b) Not being able to comprehend or comply with instructions.

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2004-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
walking velocity | six months

SECONDARY OUTCOMES:
Energy expenditure index | six months

CONTACTS AND LOCATIONS:
Overall Officials: Yeshayahu Hutzler, Ph.D, Study Director — Israel Sport Center for the Disabled
Locations (1):
- Israel Sport Center for the Disabled, Ramat Gan, Israel